CLINICAL TRIAL: NCT00142974
Title: Assessment of the Effect of Tegaserod (2 mg Tid and 6 mg Tid) on Dyspeptic Symptoms in Diabetic Patients With Symptoms of Diabetic Gastropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early in April 2005 due to low patient enrollment
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CHTF919G2203
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Diabetic Gastropathy
Keywords: Diabetes, tegaserod, gastropathy
MeSH Terms: conditions — Diabetes Mellitus; Stomach Diseases | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
This study is being done to evaluate the safety, tolerability and satisfactory relief of tegaserod against dyspeptic symptoms in diabetic patients with symptoms of diabetic gastropathy.

ELIGIBILITY:
Inclusion Criteria:

* History of Type 1 or insulin-requiring Type 2 diabetes for at least 3 years
* GI symptoms for at least 2 months before entering study

Exclusion Criteria:

* Very high body weight
* Significant diarrhea
* Ulcers

Symptom severity score collected via diary Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-05; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Reduction in weekly mean of a daily composite diabetic gastropathy dyspeptic symptom severity score throughout 6 weeks of treatment.

SECONDARY OUTCOMES:
Weekly global measure of dyspeptic symptom relief.
Weekly mean severity of individual dyspeptic symptoms (nausea, vomiting, retching, epigastric/stomach, discomfort/pain, postprandial fullness, bloating, early satiety).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Basel
Locations (1):
- Novartis, Basel, Switzerland